CLINICAL TRIAL: NCT00402571
Title: Assessment of Hepatic Function in Alcoholic Patients Administered Therapeutic Dosing of Acetaminophen- a Multicenter Study
Brief Title: Hepatic Function During and Following Three Days of Acetaminophen Dosing in Alcoholics
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Denver Health and Hospital Authority (Other)
Collaborators: McNeil Consumer & Specialty Pharmaceuticals, a Division of McNeil-PPC, Inc. (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double
Other Study IDs: COMIRB #00-715
Record Dates: First submitted 2006-11-20; First posted 2006-11-22 (Estimated); Last update posted 2009-02-09 (Estimated); Status verified 2009-02

CONDITIONS: Alcohol Related Disorders
Keywords: acetaminophen; alcohol; liver injury
MeSH Terms: conditions — Alcohol-Related Disorders | interventions — Acetaminophen

INTERVENTIONS:
Drug: acetaminophen

SUMMARY:
The study objective was to determine whether liver injury develops in alcoholic patients who ingest therapeutic doses of APAP for three consecutive days. Volunteers were recruited from two community detoxification centers to take either acetaminophen (4 g/day) or placebo for 3 consecutive days and remain in the facility an additional 2 days for monitoring. The primary measures were aminotransferase measures taken at baseline and Days 2-5. We hypothesized that there would be no difference in aminotransferase measures between the acetaminophen and placebo study groups.

ELIGIBILITY:
Inclusion Criteria

Any patient, regardless of gender or ethnicity, who was:

1. 18 years or older
2. admitted to one of the two controlled access alcohol detoxification centers with a positive BAL at the time of admittance
3. signed a written informed consent form.

Patients were excluded from the study at baseline if any of the following were present:

1. serum acetaminophen level greater than 20 mcg/ml
2. serum AST or ALT levels greater than 200 IU/L
3. INR greater than 1.5
4. if female, positive for beta-subunit of chorionic gonadotropin
5. clinically intoxicated, psychiatrically impaired or unable to give informed consent
6. known hypersensitivity to acetaminophen
7. history of ingesting more than four grams of APAP per day for any of the four days preceding study enrollment
8. currently enrolled in another trial or had been enrolled in another trial in the preceding three months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 420
Dates: Start 2002-01; Study Completion 2004-07

PRIMARY OUTCOMES:
mean change in serum aminotransferase levels between study groups

SECONDARY OUTCOMES:
proportion of subjects tht developed an abnormal aminotransferase level
proportion of subjects that developed hepatotoxicity (ALT>1000 IU/L)
proportion of subjects that developed drug induced liver injury

CONTACTS AND LOCATIONS:
Overall Officials: Richard C Dart, MD, PhD, Principal Investigator — Denver Health/Rocky Mountain Poison & Drug Center
Locations (2):
- United States (2):
  - Denver CARES, Denver, Colorado
  - Recovery Centers of King County, Seattle, Washington